CLINICAL TRIAL: NCT00313495
Title: Cooperative Huntington's Observational Research Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HP Therapeutics Foundation (Other)
Collaborators: Huntington Study Group (Network)
Responsible Party: Ira Shoulson, MD/Principal Investigator, University of Rochester
Other Study IDs: COHORT
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Huntington Disease
Keywords: Huntington disease, observational, family members, biomarker
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, DNA and Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect prospective data from individuals who are part of a Huntington Disease (HD) family, in order to relate phenotypes between individuals and families with each other and genetic factors in order to learn more about HD, develop potential treatments for HD, and to plan for future research studies of experimental drugs aimed at slowing or postponing the onset and progression of HD.

DETAILED DESCRIPTION:
COHORT (Cooperative Huntington Observational Research Trial) is a coordinated research effort by Huntington Study Group research centers worldwide to prospectively collect data from consenting individuals who are affected by Huntington's disease (HD) and who are part of an HD family. The systematically accrued data from annual prospective assessments will relate clinical characteristics (phenotypes) between families with genetic and environmental factors. The knowledge from these relationships will better inform us about the onset and progression of HD, help identify potential interventions for HD, and aid in planning research studies of experimental treatments aimed at slowing or postponing the onset of HD. The consented collection of biological samples will further provide research material and correlative data for scientists to identify biomarkers that parallel the development and progression of HD. Identification of biomarkers will in turn contribute to our understanding of HD and enhance the efficiency and power of disease-modifying therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* (1) MANIFEST/PRE-MANIFEST HD: Individuals of any age who are affected by HD OR an individual 18 years or older who - has tested positive for the HD gene.
* (2) INDIVIDUALS AT RISK: An individual 18 years or older who has not undergone DNA testing for the mutation responsible for HD and who is a first degree relative (parent, sibling, child) of an individual with Manifest or pre-manifest HD OR an older adolescent 15 to 17 years of age who has a parent with manifest HD or pre-manifest HD enrolled in COHORT.
* (3) ADULTS AT SECONDARY RISK: An individual 18 years of age or older who has not undergone DNA testing for the mutation responsible for HD and is a grandparent or grandchild of an individual enrolled in COHORT who has manifest HD or pre-manifest HD
* (4) CONTROL: A spouse or caregiver, 18 years of age or older, of an individual enrolled in COHORT who has manifest HD or pre-manifest HD
* (5) ADULT GENE NEGATIVE: An individual, 18 years of age or older, with a family history of HD who has undergone DNA testing and does not carry the genetic mutation responsible for HD.

Exclusion Criteria:

* (1) Anyone who does not fit the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. An individual of any age that is affected by Huntington's disease
  2. An individual 18 years of age or older, who has tested positive for the HD gene
  3. An individual 18 years of age or older who is a parent, sibling or child of an individual affected by HD
  4. An older adolescent 15 to 17 years of age, who has a parent affected by HD enrolled in COHORT, or a parent who has tested positive for the HD gene enrolled in COHORT (at select sites)
  5. Grandparents and grandchildren of anyone participating in COHORT who fulfills the requirements of (the above) category (1) or (2)
  6. HD family members who have no risk for HD due to no family history (spouses or caregivers)
  7. HD family members who have undergone DNA testing and does not carry the genetic mutation responsible for HD.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shoulson, MD, Principal Investigator — University of Rochester/Huntington Study Group
Locations (52):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Colorado Neurological Institute, Littleton, Colorado
  - University of Connecticut, Hartford, Connecticut
  - Institutue for Neurodegenerative Disorders, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hereditary Neurological Disease Center, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee-Memphis, Memphis, Tennessee
  - Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Booth Gardner Parkinsons Center, Kirkland, Washington
- Australia (3):
  - Westmead Hospital, Wentworthville, New South Wales
  - The University of Melbourne, Kew, Victoria
  - Graylands, Selby-Lemnos & Special Care Health Services, Perth, Western Australia
- Canada (8):
  - University of Calgary Medical Clinic, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Movement Disorder Clinic Deer Lodge Centre, Winnipeg, Manitoba
  - Movement Disorders Clinic, Deer Lodge Centre, Winnipeg, Manitoba
  - Halifax Infirmary, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - The Centre for Addiction and Mental Health, Markham, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec

REFERENCES:
- [Derived] Connors MH, Teixeira-Pinto A, Loy CT. Psychosis and longitudinal outcomes in Huntington disease: the COHORT Study. J Neurol Neurosurg Psychiatry. 2020 Jan;91(1):15-20. doi: 10.1136/jnnp-2019-320646. Epub 2019 Oct 13. PMID 31611263
- [Derived] Dorsey ER, Beck CA, Darwin K, Nichols P, Brocht AF, Biglan KM, Shoulson I; Huntington Study Group COHORT Investigators. Natural history of Huntington disease. JAMA Neurol. 2013 Dec;70(12):1520-30. doi: 10.1001/jamaneurol.2013.4408. PMID 24126537
- [Derived] Huntington Study Group COHORT Investigators; Dorsey E. Characterization of a large group of individuals with huntington disease and their relatives enrolled in the COHORT study. PLoS One. 2012;7(2):e29522. doi: 10.1371/journal.pone.0029522. Epub 2012 Feb 16. PMID 22359536
- See also: The Huntington Study Group (HSG) is a non-profit group of physicians and other health care providers from medical centers in the U.S., Canada, Europe and Australia, experienced in the care of Huntington patients and dedicated to clinical research of HD. — http://www.Huntington-Study-Group.org